CLINICAL TRIAL: NCT01196039
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy, Safety, and Tolerability of Intravenous MEMP1972A in the Prevention of Allergen-Induced Airway Obstruction in Patients With Mild Asthma
Brief Title: A Study of MEMP1972A in the Prevention of Allergen-Induced Airway Obstruction in Patients With Mild Asthma (SOLARIO)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MOP4843g; GA01332 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2010-09-03; First posted 2010-09-08 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Experimental)
  Interventions: Drug: MEMP1972A
- B (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: MEMP1972A — Intravenous repeating dose
  Arms: A
Drug: placebo — Intravenous repeating dose
  Arms: B

SUMMARY:
This Phase II, double-blind, placebo-controlled, randomized, parallel-group study is designed to evaluate the efficacy, safety and tolerability of MEMP1972A when administered to patients by intravenous (IV) infusion for the treatment of allergen-induced asthma.

ELIGIBILITY:
Inclusion Criteria:

* Mild, stable allergic asthma
* History of episodic wheeze and shortness of breath
* FEV1 at baseline >= 70% of the predicted value
* Males or females who are surgically sterilized, post menopausal for the past year, or are using two acceptable methods of contraception against pregnancy through at least 5 months following the last administration of study drug
* Documented PC20 value for prediction of the starting allergen concentration at screening
* Positive skin prick test to common standard aeroallergens extracts
* Positive allergen-induced early and late airway response

Exclusion Criteria:

* A worsening of asthma within 6 weeks preceding Visit 1
* Acute respiratory infection within 6 weeks preceding Visit 2 or any ongoing chronic infection
* History of recurrent bacterial infection as an adult or history or presence of any chronic infectious condition
* Risk of exposure, as determined by the investigator, to water-borne parasites or clinical diagnosis of parasitic infection that is untreated within 3 months prior to Visit 5
* Lung disease other than mild allergic asthma
* History of clinically significant hypotensive episodes or symptoms of fainting, dizziness, or lightheadedness
* History or symptoms of cardiovascular disease
* History or symptoms of significant neurologic disease
* History of significant hepatic or renal impairment
* Evidence of an active or suspected cancer or history of treatment for cancer
* History or symptoms of clinically significant autoimmune disease
* Any acquired or congenital immune deficiency
* Confirmed positive test for HIV or hepatitis B or C
* Concomitant disease or condition, which could interfere with the conduct of the study, or for which the treatment might interfere with the conduct of the study, or which would, in the opinion of the investigator, poses an unacceptable risk to the patients in this study
* History of serious adverse reaction or hypersensitivity to any drug
* Clinically significant abnormal chest radiograph within the last 12 months
* Pregnancy or lactation or positive serum pregnancy test at screening
* Use of corticosteroids, immunosuppressives, anticoagulants, or any medications that may interact with study drug within 4 weeks prior to Visit 2
* Chronic use of any other medication for treatment of allergic lung disease other than short-acting Î²2-agonists or ipratropium bromide
* Use of cromoglycate, nedocromil, leukotriene receptor antagonists, and inhibitors of 5-lipoxygenase are not permitted within 4 weeks prior to Visit 2
* Allergen or peptide immunotherapy within 6 months prior to study treatment
* Participation in any other investigational drug study within the preceding 30 days or 5 half-lives of that drug, whichever is longer at the time of Visit 2
* Current (or history of) treatment with a monoclonal antibody or chimeric biomolecule within the past 5 months, including omalizumab, at the time of Visit 2
* Use of statins are not permitted within 4 weeks prior to Visit 2
* Received live or attenuated vaccine within 30 days prior to Visit 5
* Regular use of tobacco products of any kind or within the previous 6 months, or smoking history > 10 pack-years
* History of drug or alcohol abuse
* Donation of blood over 500 mL within 3 months prior to Visit 5
* Unwillingness or inability to comply with the study protocol for any other reason

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-12; Primary Completion 2011-08 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Late airway response (LAR) area under the concentration-time curve (AUC) (percent decline in forced expiratory volume in 1 second [FEV1] over time) | Between 3 and 7 hours after allergen challenge at Day 86 after the first dose

SECONDARY OUTCOMES:
Maximum percent decline in FEV1 | Immediately prior to the allergen challenge to between 3 and 7 hours after allergen challenge on Day 86 after the first dose
Change in methacholine challenge PC20 relative to the pre-allergen challenge PC20 | Day 87
Maximum percent decline in FEV1 and early airway response (EAR) AUC (percent decline in FEV1 over time) | Between 0 and 3 hours after post-treatment allergen challenge

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Harris, MD, Ph.D, Study Director — Genentech, Inc.
Locations (7):
- Canada (6):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Hamilton, Ontario
  - Ste. Foy, Quebec
  - Saskatoon, Saskatchewan
- Stockholm, Sweden

REFERENCES:
- [Derived] Gauvreau GM, Harris JM, Boulet LP, Scheerens H, Fitzgerald JM, Putnam WS, Cockcroft DW, Davis BE, Leigh R, Zheng Y, Dahlen B, Wang Y, Maciuca R, Mayers I, Liao XC, Wu LC, Matthews JG, O'Byrne PM. Targeting membrane-expressed IgE B cell receptor with an antibody to the M1 prime epitope reduces IgE production. Sci Transl Med. 2014 Jul 2;6(243):243ra85. doi: 10.1126/scitranslmed.3008961. PMID 24990880